CLINICAL TRIAL: NCT07221409
Title: Pilot Study to Assess Safety, Tolerability and Efficacy of Virtual Reality in Cancer Patients
Brief Title: Virtual Reality Intervention to Improve Psychological Symptom Burden for Cancer Patients Undergoing Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-002609; NCI-2025-07303 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25-002609 (Other: Mayo Clinic in Florida)
Record Dates: First submitted 2025-09-29; First posted 2025-10-27 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Adjustment Disorder; Anxiety Disorder; Depression; Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm; Cancer
Keywords: Virtual Reality Therapy; VR Therapy; Non-Pharmacologic Intervention; Cancer Supportive Care
MeSH Terms: conditions — Adjustment Disorders; Anxiety Disorders; Depression; Neoplasms | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality (VR) Headset Intervention (Experimental): Participants will undergo a single VR session to assess feasibility, tolerability, and changes in anxiety, depression, and fatigue.
  Interventions: Other: Questionnaire Administration; Other: Virtual Reality (VR) Intervention

INTERVENTIONS:
Other: Questionnaire Administration — Participants will complete pre- and post-intervention questionnaires to assess symptoms of anxiety, depression, and fatigue.
Other: Virtual Reality (VR) Intervention — Participants will engage in a single-session immersive Virtual Reality (VR) experience lasting approximately 20-30 minutes. The VR content will include calming, guided experiences such as nature scenes, meditation, or breathing exercises designed to promote relaxation and reduce psychological distress. The intervention will be administered in a clinical setting.
  Other Names: VR Intervention; Virtual Technology; VR Headset

SUMMARY:
This clinical trial tests the safety, tolerability, and effectiveness of a virtual reality intervention to improve psychological symptom burden for cancer patients undergoing treatment. Virtual reality (VR) is a technology that allows users to experience and interact with three-dimensional, computer-generated environments that simulate the real world or imagined settings. The VR intervention consists of a preloaded with immersive environments designed to engage the senses through simulated sights and sounds. This may include a walk through of a serene forest, exploring vibrant coral reefs, swimming with dolphins, or standing at the base of a majestic waterfall. These environments are created to provide a relaxing and engaging experience. Completing the VR intervention may be a safe and effective way to improve quality of life, reduce anxiety, enhance focus, and promote healthy living for cancer patients undergoing treatment.

ELIGIBILITY:
Inclusion Criteria:

* History of cancer
* Age between 18 to 90 years
* Undergoing in-patient chemotherapy, bone marrow transplant (BMT), chimeric antigen receptor (CAR)-t, & out-patient chemotherapy

Exclusion Criteria:

* History of bipolar disorder, major depression, bipolar disorder, anxiety disorder, post traumatic stress disorder (PTSD), obsessive compulsive disorder (OCD), psychotic disorder, schizophrenia, personality disorder, substance use disorder other than caffeine or tobacco. History of suicidal ideation or attempt
* History of treatment resistant depression, psychiatric hospitalization, syncope, transient ischemic attack (TIA), stroke, epilepsy, electroconvulsive therapy, benign positional vertigo, Meniere's disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2027-10-08 (Estimated); Study Completion 2027-10-08 (Estimated)

PRIMARY OUTCOMES:
Successfully complete the virtual reality (VR) intervention (Feasibility) | Baseline
  Feasibility of VR will be assessed by the proportion of participants who successfully complete the intervention.
Absence of major issues during administration (Feasibility) | Baseline
  Feasibility of VR will be evaluated by the absence of (low/no recorded incidence of) major technical or usability issues during administration
Acceptability | Baseline
  Will be assessed via the Post-Study Exit Interview Questionnaire, a questionnaire developed specifically for this study. It consists of 17 questions. Eight questions relate to the VR experience (e.g., comfort of headset, control of actions in VR environment, understandability of instructions, technical issues). Five questions relate to symptoms (e.g., dizziness, nausea, headache) or discomfort experienced during and immediately following VR use. The remaining questions relate to helpfulness of intervention, improvement suggestions, other feedback, and interest in learning more about services and resources. Results will be analyzed descriptively.

SECONDARY OUTCOMES:
Change in anxiety | Baseline (pre- to post-intervention, approximately 1.5 hours)
  Assessed using the Patient Reported Outcome Measurement Information System (PROMIS) Cancer Bank v1.0 - Anxiety scale, which is specifically designed to measure anxiety in cancer patients. The scale consists of 22 questions related to anxiety symptoms over the past 7 days. Questions are answered on a 5-point scale (Never, Rarely, Sometimes, Often, Never). Higher scores reflect greater levels of anxiety.
Change in depression | Baseline (pre- to post-intervention, approximately 1.5 hours)
  Assessed using the PROMIS Cancer Bank v1.0 - Depression scale, which measures depressive symptoms in individuals with cancer through self-reported questions. The scale consists of 30 questions related to emotional distress over the past 7 days. Questions are answered on a 5-point scale (Never, Rarely, Sometimes, Often, Never). Higher scores indicate greater emotional distress (depression).
Change in fatigue | Baseline (pre- to post-intervention, approximately 1.5 hours)
  Assessed using the PROMIS Cancer Bank v1.0 - Fatigue scale, which measures experience of fatigue (frequency, duration, intensity) over the past 7 days and its impact on physical, mental, and social activities. The scale consists of 54 questions answered on a 5-point scale such as Not at all, A little bit, Somewhat, Quite a bit, Very much or Never, Rarely, Sometimes, Often, Always. Higher scores indicate greater fatigue.
Change in overall quality of life | Baseline (pre- to post-intervention, approximately 1.5 hours)
  Assessed via Uniscale questionnaire, which consists of a single question assessing overall quality of life during the past week. The question is answered on a 10-point Likert scale where 0=As bad as it cand be and 10=As good as it can be.

CONTACTS AND LOCATIONS:
Overall Officials: Juan C. Cardenas Rosales, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials